CLINICAL TRIAL: NCT03138460
Title: Effect of New Pain Modulating Substances in Orthopedics
Brief Title: Analysis of Orthopedic Patients Response to New Pain Modulating Substances and Drugs
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, DROR ROBINSON, Head Orthopedic Research Unit, Rabin Medical Center
Other Study IDs: 0612-16
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard medications crossed over to cannabis

SUMMARY:
Data of patient reported outcomes (PRO) are collected during treatment with various pain alleviation methods (drugs or substances)

DETAILED DESCRIPTION:
The study aims at collecting BPI (brief pain inventory) and other PRO of patients in need of pain relief due to chronic orthopedic pain conditions

ELIGIBILITY:
Inclusion Criteria:

Chronic pain of orthopedic origin treated for at least one year unsuccessfully

Exclusion Criteria:

contra-indication for cannabis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic pain sufferers mostly low back pain but also fibromyalgia and arthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Brief pain inventory score (BPI) | 2 years
  score of PRO

CONTACTS AND LOCATIONS:
Overall Officials: dror robinson, md, Principal Investigator — head orthopedic research unit
Locations (1):
- Hasharon Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No